

## **Informed Consent**

Analysis of the Safety and Efficacy of Administering Umbilical Cord Mesenchymal Stem Cell Secretome in Patients With Severe Erectile Dysfunction Non-responsive to Sildenafil

Date: 6 October 2025



## INFORMED CONSENT FORM Principal Investigator : Dr. dr. Ria Margiana, Sp.And, M.Biomed Information Provider Information Recipient Name Birthdate (Age) Gender Address Phone TYPE OF CONTENT **MARK INFORMATION** 1. Research Title Comparative Analysis of Safety and Efficacy between Administration of Secretome and Exosomes from Umbilical Cord-Derived Mesenchymal Stem Cells in Patients with Erectile Dysfunction 2. Research The aim of this study was to analyze the differences in safety (local bleeding, hematoma, infection, pain) and Purpose efficacy after administering umbilical cord mesenchymal stem cell secretome and exosomes to patients with Erectile Dysfunction. This is an experimental study, assessing pre- and 3. Research Methodology post-test scores. Patients who consent to the study will undergo an intracavernous injection of secretome/exosomes. Follow-up will be conducted at 2 weeks and 1 month after the study to evaluate several safety and efficacy parameters of the secretome/exosomes. 4. Risks and Side Secretomes and exosomes have been used as adjuvant therapy and have not caused significant side Effects in Research effects. However, bleeding, bruising, tenderness, and swelling can occur in some individuals. During the study, researchers prepared the necessary safeguards in case of any adverse events. This protection included consultation and hospitalization services for potential side effects following the intervention. If bleeding, bruising, tenderness, and swelling occurred, subjects were informed beforehand to immediately apply a cold compress, which could be applied with cold water or ice cubes, for 10-20 minutes. If swelling occurred, a steroid injection was



| 5. | Benefits of | given. If localized urticaria occurred, a topical antihistamine was given. If symptoms persisted and were accompanied by fever, the researchers and the hospital where the study was conducted would administer treatment in accordance with applicable Clinical Practice Guidelines, at the researchers' expense. The benefits you can get include receiving adjuvant |
|---|---|---|
| | research include<br>benefits for<br>research<br>subjects | therapy for erectile dysfunction using UC-MSC secretome or exosomes and understanding its effects on your erectile function. |
| 6. | Research Procedures (written in detail using layman's language) | 1. You will be interviewed by a doctor who will ask about your name, age, medical history, sexual history, medication history, allergies, smoking habits, and drinking habits. 2. You will undergo a physical examination by a doctor to assess your health and sexual health. 3. Before the injection therapy, you will be informed about the effectiveness and possible complications of the treatment and will complete several initial questionnaires for parameters [International Index of Erectile Function-5 (IIEF-5), Erectile Hardness Score (EHS), and Nocturnal Penile Tumescence (NPT)]. 4. On the day the study begins, you will be asked to come in for the interventional procedure. 5. The injection of stem cell-derived substances (UC-MSC secretome or exosomes) into the penis (intracavernosa) will be performed by a qualified doctor. The UC-MSC secretome used is a product developed by PT Kalbe. 6. You will be injected with 0.5 mL of UC-MSC secretome/exosomes into the penis (intracavernosa) using a 30-gauge needle according to a sterile protocol. Equal volumes are administered on both sides of the penile shaft, totaling 1 mL. The injections are given twice daily, on both sides of the penile shaft. 7. Tolerability is assessed by observing and questioning the subjects regarding pain during the intracavernosal injection. Pain intensity is rated on a visual analog scale of 0-10, where 0-3 represents mild pain, 4-6 represents moderate pain, and 7-10 represents severe pain. 8. After the injection, the |



| 7. | Discomfort of research subjects | safety of the secretome will be assessed by examining the injection site for signs of bleeding, bruising, tenderness, swelling, coldness (hypothermia), heat (hyperthermia), redness (erythema), hives (urticaria), or fluid-filled hives (induration). Vital signs (temperature, heart rate, respiratory rate, and blood pressure) will be measured. You will also be interviewed for other possible side effects. The safety of the therapy will be assessed immediately, 24 hours after injection, and 1 month after injection through a physical examination. 9. The effects of intracavernous injection therapy will be assessed qualitatively using the International Index of Erectile Function-5 (IIEF-5), Erectile Hardness Score (EHS), and Nocturnal Penile Tumescence (NPT) questionnaires at baseline, 1 month, and 6 months after the intervention. 10. Patients will continue to receive their primary therapy, oral sildenafil. Discomfort may occur during intracavernous injections, but they will be administered by qualified medical personnel. After the injection, redness, | |
|---|---|---|---|
| | (potential | bleeding, infection, and fever may occur. | |
| | discomfort) | | |
| 8. | Alternatif penanganan | The researchers provided consultation and hospital care for potential side effects following the intervention. Subjects were instructed to immediately apply a cold compress, typically with cold water or ice cubes, for 10–20 minutes, as first aid. If swelling persisted, a steroid injection was administered. If localized hives occurred, topical antihistamines were administered. If symptoms persisted and fever developed, the researchers and the hospital where the study was conducted would administer treatment in accordance with the applicable Clinical Practice Guidelines, with the researcher responsible for the costs. | |
| 9. | Maintaining data confidentiality | All data collected in this study will be kept confidential. Presentations of research results at scientific meetings/conferences and publications in scientific journals will not include your name. However, ethics committees and national regulatory bodies regulating the use of medicines will have access to the research data for verification. | |
| LSubj | ect Initial | informed con | sent_RSUI |



| NRM | : | 1 |
|------------|---|---|
| Name | : | |
| Gender | : | |
| Birth date | : | |

| 10 | Componentian if | If the complaint does not improve and is commented |
|---|---|---|
| 10. | Compensation if | If the complaint does not improve and is accompanied |
| | side effects | by fever, the researcher and the hospital where the |
| | occur | research is taking place will carry out management in |
| | | accordance with the applicable Clinical Practice |
| | | Guidelines, with costs borne by the researcher. |
| 11. | Name and | Dr. dr. Ria Margiana, Sp.And, M.Biomed |
| | address of | Perumahan Taman Tanah Baru B2 no. 7, Tanah Baru, |
| | researcher and | Beji, Depok |
| | contact | +62 811-1775-515 |
| | telephone | |
| | number | |
| 12. | Number of | 12 person |
| | subjects | |
| 13. | Potential danger | In general, this study did not cause significant side |
| | | effects, but in some people bleeding, bruising, |
| | | tenderness, and swelling may occur. |
| 14. | Costs incurred | None |
| 15. | Incentives for | Rp300.000 |
| | subjects | |

| After reading the explanation | on pages 1 to 4 regarding the research to be conducted |
|---|---|
| by entitled "Comp | parative Analysis of the Safety and Efficacy of Administering |
| Secretome and Exosomes from | n Umbilical Cord-Derived Mesenchymal Stem Cells to Patients |
| with Erectile Dysfunction," I have | e fully understood this information. |
| By signing this form, I agree to | o participate in the above research voluntarily without coercior |
| from any party. If at any time I | feel I have been harmed in any way, I have the right to withdraw |
| this consent. | |
| Signature | Date |
| Name | |
| Guardian Signature | Date |
| Guardian Signature | |
| Subject Initial | informed consent_RSUI |



| NRM | : | ) |
|------------|---|---|
| Name | : | |
| Gender | : | |
| Birth date | : | |
| | | ) |

I have explained to the subject correctly and honestly the purpose of the research, the benefits of the research, the research procedures, as well as the potential risks and discomforts that may arise (a detailed explanation in accordance with the things I marked above. I have also answered questions related to the research to the best of my ability.

| Researcher Signature | <del></del> |
|----------------------|-------------|
| · · | Date |
| Researcher Name | |